CLINICAL TRIAL: NCT06921278
Title: Psychometric Development of the Alcohol and Drug Respiratory Health Questionnaire and Evaluation of a Lung Health Clinic
Brief Title: Development of the Drug and Alcohol Respiratory Health Test
Acronym: DARHT
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: DARHT
Record Dates: First submitted 2025-03-21; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Disease; Substance-Related Disorders; COPD; Asthma; Lung Cancer; Tuberculosis; Bronchitis; Pneumonia; Obstructive Sleep Apnea
MeSH Terms: conditions — Respiration Disorders; Substance-Related Disorders; Pulmonary Disease, Chronic Obstructive; Asthma; Lung Neoplasms; Tuberculosis; Bronchitis; Pneumonia; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this study is to develop a brief Drug and Alcohol Respiratory Health Test (DARHT) and offer it for routine use in clinical assessment and medical reviews

DETAILED DESCRIPTION:
Respiratory diseases are highly prevalent among adults with substance use disorder. Inhaling drugs are risk factors, and cigarette smoking contributes to 90% of COPD cases. The substance use disorders population faces barriers to accessing healthcare, leading to under-diagnosis and including stigma, exacerbating the unmet need for effective respiratory disease management. There is no population-specific screening instrument in NHS and Third Sector addiction services. The lack of a validated screening tool means Respiratory health symptoms may be overlooked or attributed to other causes. The aim of this trial is to develop a brief Drug and Alcohol Respiratory Health Test (DARHT) and make it available for clinical assessment and medical reviews. The primary research question is to determine if the DARHT achieves satisfactory diagnostic accuracy with gold-standard spirometry. The study will be open to any enrolled adult (age >18 years) patients at our treatment clinic (NHS secondary care) who reports inhaling (smoking) tobacco, cannabis, cocaine, opioids, or consuming alcohol in the past 28 days. Volunteer and informed and consenting participants will be invited to: (1) complete a brief study questionnaire that includes the DARHT, then take a spirometry and pulse oximetry test; (2) return to the clinic after 3-7 day to complete the DARHT with a different interviewer. Participants with a positive case evaluation on the DARHT or spirometer will be referred to primary or specialist services. The investigators will contact participants referred after 6 weeks to determine their progress and the PHQ-4 and EQ-5D-L to evaluate changes in quality of life. The first 20 participants referred to specialist care will be invited to a Lung Health Clinic where the investigators will offer a psycho-social intervention for advice and support.

ELIGIBILITY:
Inclusion Criteria:

1. >18 (no upper age limit)
2. Inhalation (smoking) of tobacco, or cannabis, or cocaine, or opioids, or use of alcohol in the past 28 days
3. Possession of a personal mobile phone to arrange follow-up appointments

Exclusion Criteria:

1. Reported physical health condition that would mean spirometry contra-indicated - including heart attack, unstable angina, pulmonary embolism,
2. Reported surgery in the past 3 months for an eye, chest, or abdominal condition that would mean spirometry contra-indicated
3. Likely inability to complete study due to criminal justice involvement with legal proceedings risking incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Addictions Community Centre for those suffering from substance-related disorders who may also have underlying respiratory diseases.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-11-11 (Estimated); Study Completion 2025-11-11 (Estimated)

PRIMARY OUTCOMES:
A brief respiratory health screening questionnaire | Day 1 and Day 3-7
  To investigate the accuracy of a brief respiratory health screening questionnaire in highlighting respiratory health symptoms in participants with Substance Use Disorders.

SECONDARY OUTCOMES:
Specialist nurse and psychology assistant delivered Lung Health Clinic | Week 1 to Week 6
  Evaluate the effectiveness of a specialist nurse and psychology assistant delivered by the Lung Health Clinic in improving respiratory health referrals, airway medication updates and adherence, service satisfaction, and quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- South London & Maudsley NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No